CLINICAL TRIAL: NCT00212446
Title: Pilot Study to Evaluate a Prototype Electronic Uterine Inhibitor to Prevent Preterm Contractions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10-173
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Preterm Birth
Keywords: Tocolysis; Electrical Pacemaker
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrical Intervention (Experimental): Electrical intervention (EI) is bipolar, constant-current (1-20 mA), square-wave pulses in 20% duty cycles. Women in preterm labor have an electrode placed vaginally; tocodynamometric contraction timing and fetal heart rate are monitored continuously. Successive 20-minute periods include pre-control period (C1); the EI period, in which a 10-second current burst is delivered at expected contraction times; and a post-EI control period (C2).
  Interventions: Device: Electrical Intervention (EI)

INTERVENTIONS:
Device: Electrical Intervention (EI) — Electrical intervention (EI) is bipolar, constant-current (1-20 mA), square-wave pulses in 20% duty cycles. Women in preterm labor have an electrode placed vaginally; tocodynamometric contraction timing and fetal heart rate are monitored continuously. Successive 20-minute periods include pre-control period (C1); the EI period, in which a 10-second current burst is delivered at expected contraction times; and a post-EI control period (C2).

SUMMARY:
Use an electrical-inhibition (EI)/uterine pacemaker device similar to an electrical heart pacemaker to deliver a weak electrical current to the human uterus that will rapidly and safely inhibit the unwanted premature uterine contractions of preterm birth.

DETAILED DESCRIPTION:
The preterm birth rate in the United states has been stubbornly stuck at 10.5% or higher since the 1950's. The 2011 rate, 11.72%, is the most recent level available. That comes to about a half a million preterm births per year in the United States alone.

Premature birth and the attendant complications are among the greatest health problems in the world today and contribute to about 85% of all neonatal deaths, that is, deaths of infants from the time of birth until1 month old.

During the past ten years, there has been developed a novel method to effectively and objectively inhibit uterine contractility during the birthing process.

The method is nonpharmaceutical, and thus, avoids systemic side effects and has the potential to be noninvasive and easy to master.

This method uses an electrical intervention (EI)/uterine pacemaker device that will allow for rapid and reversible inhibition of preterm uterine contractions and preterm birth.

The following is a brief account of the electrical properties of the myometrium and why these properties may be affected by electrical intervention (EI).

The contractile activity of the uterus is a direct consequence of the underlying electrical activity in the myometrial cells. The sequence of contraction and relaxation of the myometrium results from the cyclic depolarization and repolarization of the membranes of the muscle cells.

The uterus at term has been shown to be myogenic just like the heart. The uterus will contract spontaneously without neuronal control, like the heart, and form gap junctions interconnecting the cells just like the syncytium of the heart. Also, both are excitable tissues with similar current flows.

Electrical Intervention (EI) has successfully inhibited myometrial or uterine contractions in many different species e.g. sheep, rabbit, rat, and human (in vitro). The EI was effective in live animals when used on the uterus either directly attached or transvaginally.

The electrical pacemaker (Inch Inc., Brooklyn, NY) used in this work is a self-contained portable device with integrated circuits, housed in a box about eight inches on all sides. EI is delivered as 10-second bursts of bipolar, constant-current, square-wave pulses in 20% duty cycles. A 20% duty cycle consists of a pulse of current at the given amperage lasting 20% of the cycle, followed by a period without current for the remaining 80% of the cycle. The number of cycles per second defines the frequency in Hertz (Hz). Because the duty cycle is constant at 20%, a 10-second burst always delivers current for a total of 2 seconds, with the frequency determining the length and number of individual pulses, in milliseconds (msec), during the burst.

Participants were enrolled beginning in February 2005. IRB approval was in place at New York Downtown Hospital, Manhattan, NY, from inception until March 2013, when it ceased to be a study site. During the study period at Downtown Hospital, 3 participants overall were enrolled and studied. St. Luke's Roosevelt Hospital Center, Manhattan, NY, became a study site when it received IRB approval in January 2010 and at present is the only study site, and has continuing IRB approval. While under IRB approval, 5 patients have been enrolled and studied at St. Luke's and Roosevelt. Each participant has given written informed consent. To date, 53 women have been recruited overall, and 8 have given informed consent and been studied.

Those studied are females 18 years old or older, between 24-34 weeks gestation, have a reassuring fetal heart rate (FHR) tracing, and in preterm labor as defined by the American College of Obstetrics and Gynecology (ACOG). The participants must have persistent uterine contractions, with 4 every 20 minutes or 8 every 60 minutes, and any one or more of the following: documented cervical change, > 1 cm cervical dilation, or > 80% cervical effacement. The exclusion criteria are the same as for most tocolytic therapy; most importantly, premature rupture of the membranes (PROM), and additionally, severe preeclampsia, severe abruption placenta, chorioamnionitis, fetal death, fetal anomaly incompatible with life, severe fetal growth restriction or estimated fetal weight (EFW) <5%, mature fetal lung studies, maternal cardiac arrhythmias, a permanent cardiac pacemaker, a fetal cardiac arrhythmia, or any other contraindication for tocolysis.

The women have a pacemaker electrode placed vaginally. A 5 (1.67mm) or 6 (2.00mm) French electrode catheter with distal 4x2mm platinum alloy rings 5mm apart (C. R. Bard, Inc., Lowell, MA, USA) is manually placed into the posterior vaginal fornix next to the external cervical os. The catheter's proximal end is taped to the patient's thigh and its connecting cable attached to the pacemaker, which can generate a weak bipolar electrical current (0-20 mA, 0-50 msec/pulse, 50 Hz). In the study, the EI current is increased slowly, as needed, up to a maximum of 17 mA.

The human study begins immediately after placing the catheter and lasts 60 minutes; FHR, uterine contraction timing, and subjective contraction amplitude are monitored during the entire study. The first 20 minutes are the control contraction period (C1). The second 20 minutes are the EI period, with a 10-second burst of current administered just prior to each expected contraction; expected contractions are determined by the timing of the C1 contractions and/or by the rise of the subjective tocodynamometer tracing above baseline levels. The third 20 minutes is the post-intervention control contraction period (C2). The contraction intervals, the times between contraction peaks (P-P), were measured in minutes for C1, EI, and C2. All statistical analyses for the human study have been performed using Statistical Analysis System (SAS) software (SAS Institute Inc., Cary, NC, USA) Version 9.2. For each period, C1, E1, and C2, the mean minutes between contractions are estimated, using the mixed-model analysis of variance (ANOVA) to account for both within-subject and between-subject variability. Pairwise differences between mixed-model ANOVA means and corresponding p-values testing for difference from zero were estimated. All hypothesis testing is performed at the 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Pending preterm birth
* vaginal birth

Exclusion Criteria:

* disease disorders including but not limited to thyroid, liver disease, HIV, diabetes or drug addiction
* using a permanent cardiac pacemaker
* have malignancies that are currently being treated or recurrent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham G Ashmead, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study period was from February 2005 through April 2012 and was performed on the labor and delivery floor of the study sites.
Period: Overall Study
Arm/Group | Electrical Intervention
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age
  years | 31.65 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Gestational Age [Mean (Standard Deviation); unit: weeks] | 31.11 (2.19)
pre-EI cervical dilatation [Mean (Standard Deviation); unit: cm] | 3.0 (2.33)
pre-EI effacement [Mean (Standard Deviation); unit: percent of effacement] | 80.00 (17.73)

OUTCOME MEASURES:

1. Primary Outcome: Uterine Contractions
Description: The first 20 minutes are the control contraction period (C1). The second 20 minutes are the EI period, with a 10-second burst of current administered just prior to each expected contraction; expected contractions are determined by the timing of the C1 contractions and/or by the rise of the subjective tocodynamometer tracing above baseline levels. The third 20 minutes is the post-intervention control contraction period (C2).
Time Frame: 20 minutes, 40 minutes, 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
minutes
  C1 | 3.18 (1.30)
  E1 | 3.78 (1.44)
  C2 | 3.20 (1.33)

2. Primary Outcome: Number of Newborn With Fetal Heart Arrhythmias
Description: Number of newborn with fetal heart arrhythmias noted
Time Frame: 60 minutes
Measure: Number; unit: newborns with fetal heart arrhythmias
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
newborns with fetal heart arrhythmias | 0

3. Secondary Outcome: Latency of Birth
Description: Latency is defined as the time from admission into hospital until birth
Time Frame: Time until delivery, up to 4 weeks
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
hours | 599.76 (56.00)

4. Secondary Outcome: Pain During the Birthing Process
Time Frame: Until birthing process is complete
Population: not collected
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Apgars Score
Description: The 1-minute score determines how well the baby tolerated the birthing process. The 5-minute score tells the health care provider how well the baby is doing outside the mother's womb.
  Five factors: Appearance (skin color), Pulse (heart rate), Grimace response (reflexes), Activity (muscle tone), Respiration (breathing rate and effort) are used to evaluate the baby's condition and each factor is scored on a scale of 0 to 2, with full scale from 0 to 10 being the best score
Time Frame: 1 minute and 5 minute after childbirth
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
units on a scale
  1 minute | 8.75 (0.71)
  5 minute | 9.0 (0.53)

6. Secondary Outcome: The Length of NICU Stay
Description: The length of Neonatal intensive care unit (NICU) stay
Time Frame: up to one month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
days | 13.42 (11.02)

7. Secondary Outcome: Gestational Age at Discharge
Description: Gestational age at discharge.
Time Frame: until after childbirth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Electrical Intervention
Number analyzed (Participants) | 8
weeks | 36.61 (2.68)

ADVERSE EVENTS:
Description: Adverse events not collected
Arm/Group | Electrical Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
it was difficult not only to obtain written informed consent from patients but also to convince their attending physicians to participate in study. Challenging to make researchers available when patients were in preterm labor and eligible for study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No